CLINICAL TRIAL: NCT03153930
Title: Metabolic Effects of Interrupting Sedentary Time in Youth In-lab and in Free-living Settings
Brief Title: Sedentary Behavior and Health Outcomes Study
Acronym: SBHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Britni Ryan Belcher, PhD, MPH, Assistant Professor of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1K01DK113062 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Lifestyle; Metabolic Disturbance; Pediatric Obesity; Physical Activity
Keywords: sedentary behavior; youth; moderating factors; metabolic outcomes
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will complete a randomized crossover study with 2 conditions: sitting continuously for 3 hours vs. interrupting sitting with 3-minute moderate intensity walking breaks every 30 minutes for 3 hours. A subset will then complete a free-living component wearing a continuous glucose monitor that will consist of habitual activity vs. interrupting periods of 30+ sedentary minutes with short activity breaks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting Only (SIT) (Placebo Comparator): In-Lab (full sample): children will sit continuously for 3 hours during an OGTT Free-living (sub-sample; N=12): children will complete their habitual sedentary behaviors over 4 days; they will also wear a continuous glucose monitor
  Interventions: Behavioral: Sitting only
- Walking Breaks (WALK) (Experimental): In-Lab (full sample): children will be asked to walk on a treadmill every 30 minutes for 3 minute bouts during a 3 hour OGTT Free-living (sub-sample; N=12): children will be prompted with an ActivPAL vtap monitor on the right thigh to perform 3-minute walking bouts whenever sedentary time has lasted longer than 30 minutes over 4 days; they will also wear a continuous glucose monitor
  Interventions: Behavioral: Walking breaks

INTERVENTIONS:
Behavioral: Walking breaks — In-Lab (full sample): participants will be asked to walk on a treadmill for 3 minutes every 30 minutes at a moderate pace during a 3-hour OGTT Free-living (sub-sample; N=12): participants will be prompted via an ActivPAL vtap monitor to walk for 3 minutes every time sedentary behavior lasts longer than 30 continuous minutes
  Other Names: Interrupting sedentary time
  Arms: Walking Breaks (WALK)
Behavioral: Sitting only — In-Lab (full sample): participants will remain seated for 3 hours during an OGTT Free-living (sub-sample; N=12): participants will perform their habitual sedentary behaviors
  Other Names: Continuous sedentary time
  Arms: Sitting Only (SIT)

SUMMARY:
This study is a randomized crossover trial to compare the effectiveness of interrupting SB on glucose homeostasis in the lab and free-living settings. All participants (N=56) will complete one screening visit to determine eligibility, complete at fitness test, and body composition analysis by bioelectrical impedance. After 7-21 days, all participants will complete two 3-hour in-lab oral glucose tolerance tests (spaced 7-21 days apart). Prior to the in-lab OGTT visits, participants will wear an activity monitor for 7 days on the right thigh. The experimental conditions for the OGTTs will be: 1) 3-hour OGTT of continuous sitting; and 2) 3-hour OGTT with sitting interrupted every 30 minutes with 3-minutes of moderate intensity walking on a treadmill. There will be a 7-21 day washout period between the OGTT visits. In addition, a subset of participants (N=12) who meet inclusion criteria and who successfully complete both OGTT visits will complete a second randomized crossover trial in the free-living environment. The experimental conditions for the free-living components will be: 1) 4 days of habitual sedentary behaviors; and 2) 4 days of prompted short exercise breaks during times in which sedentary behaviors have exceeded 30 minutes. Participants in the free-living trial will wear an activity monitor and a continuous glucose monitor.

DETAILED DESCRIPTION:
Rationale: Sedentary behavior (SB) can increase risk for type 2 diabetes. Interrupting SB is a promising strategy to reduce risk, but the long-term success is not yet clear and data on the relationship between in-lab and free-living metabolic responses are lacking. A better understanding of the relationship between metabolic responses to sitting and interrupting sitting in the lab and in a naturalistic environment will help us design effective and targeted intervention strategies to prevent type 2 diabetes in youth.

Intervention: Participants (28 healthy weight and 28 overweight/obese youth; ages 11-15 years) from an ongoing longitudinal observational study (HS-12-00446) will complete: a) an in-lab randomized crossover trial of acute metabolic responses to prolonged vs. SB interruptions; and a subset (N=12) will complete b) two 4-day continuous glucose monitoring (CGM) studies of effects of free-living habitual activity vs. SB interruptions on glucose homeostasis.

Objectives/Purpose: The overall goal is to improve metabolic outcomes by interrupting SB in youth with small bouts of exercise. The aim of this study is to investigate whether the metabolic responses to interrupting sitting are the same in a controlled lab setting and a free-living setting. This study will also try to explain why some children respond better to these short interruptions in sitting than others by using three years of physical activity, body fat, and weight trajectory data from an ongoing study (HS-12-00446).

Study Population: The study population will consist of participants currently enrolled in the Mothers and Their Children's Health (MATCH) Study (PI: Dunton; HS-12-00446; ages 11-15 years).Eligible participants will have completed 3 years of semi-annual assessments of body composition, physical activity, and dietary intake in the MATCH study.

Study Methodology: This study is a randomized crossover trial to compare the effectiveness of interrupting SB on glucose homeostasis in the lab and free-living settings. All participants (N=56) will complete one screening visit to determine eligibility, complete at fitness test, and body composition analysis by bioelectrical impedance. After 7-21 days, all participants will complete two 3-hour in-lab oral glucose tolerance tests (spaced 7-21 days apart). Prior to the in-lab OGTT visits, participants will wear an activity monitor for 7 days on the right thigh. The experimental conditions for the OGTTs will be: 1) 3-hour OGTT of continuous sitting; and 2) 3-hour OGTT with sitting interrupted every 30 minutes with 3-minutes of moderate intensity walking on a treadmill. There will be a 7-21 day washout period between the OGTT visits. In addition, a subset of participants (N=12) who meet inclusion criteria and who successfully complete both OGTT visits will complete a second randomized crossover trial in the free-living environment. The experimental conditions for the free-living components will be: 1) 4 days of habitual sedentary behaviors; and 2) 4 days of prompted short exercise breaks during times in which sedentary behaviors have exceeded 30 minutes. Participants in the free-living trial will wear an activity monitor and a continuous glucose monitor.

Study Arms: Participants will be assigned to receive in random order the continuous sitting test at the first visit and the sitting interruptions test on the second visit, or vice versa. The order of the free-living conditions will be the same as the in-lab condition order.

Endpoints/Outcomes: The primary endpoints are: insulin, C-peptide, and glucose area under the curve (AUC) in the in-lab experiments, and glucose AUC in the free-living experiments.

Follow-up: Study duration for those completing only the in-lab experiments is a minimum of 17 days and a maximum of 45 days to complete. For the subset of participants who are additionally completing the free-living component, the study duration is a minimum of 25 days and a maximum of 53 days.

Statistical Analyses: The populations for analyses include the full analytical dataset which consists of all randomized study participants, with the exception of those participants in the parent MATCH study who are not participating in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. current/past participant in the MATCH Study
2. good general health
3. fasting plasma glucose <100 mg/dL
4. BMI greater than the 5th percentile

Exclusion Criteria:

1. significant cardiac or pulmonary disease likely to or resulting in hypoxia or decreased perfusion
2. evidence of impaired glucose tolerance or type 2 diabetes
3. presence of other endocrinologic disorders leading to obesity (e.g.: Cushing Syndrome)
4. current or past anti-psychotic drugs use that would affect metabolism
5. non-diet treatment for hypertension or dyslipidemia
6. precocious puberty and/or receiving androgen and estrogen therapy
7. medication use known to affect body composition/weight

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
In-Lab: Metabolic responses | 3 hours
  glucose, insulin, and c-peptide area under the curve
Free-living: Glucose responses | 4 days
  glucose area under the curve
Predictors of in-lab glucose responses | 3 years
  Independent-sample t-tests will assess if mean in-lab glucose AUC differs within experimental condition by weight status (normal weight or overweight/obese). Independent-sample t-tests will assess if mean AUC values between conditions (delta AUC) differ by weight status. Structural equation models of latent growth curves will be used to assess the relationship between BMI z-score trajectories in the preceding 3 years, in-lab glucose AUC responses by experimental condition. Specifically, models will test if a) the higher the initial BMI z score (year 1), the higher the initial serum value (-10 min); b) the higher the initial BMI z score (year 1), the greater the change in serum AUC between experimental conditions; and c) the greater slope of the BMI z score change, the greater the change in serum AUC between experimental conditions.
Individual variations in glucose responses in-lab | 3 years
  Mixed-effects location scale models (MIXREGLS) will test how between-subject (BS) and within-subject (WS) variation in SB in the preceding 3 years are associated with glucose responses to in-lab SB interruptions. The predictors are average 3-year SB level and SB level at each year (variation in SB). The Stage 1 mixed-effects location scale model will examine random effects of between-subject variance (i.e., location) and of within-subject variance (i.e., scale), sex, baseline percent body fat, and baseline age. The Stage 2 model will assess how these variance sources from Stage 1 affect the delta AUC between in-lab prolonged SB and SB interruptions with regards to glucose (the WS effects).

SECONDARY OUTCOMES:
Relationship between in-lab and free-living glucose AUC | 5 days
  We will assess bivariate correlations between the in-lab glucose AUC and the first day of in-field glucose AUC. Linear regression will be used to estimate associations between in-lab glucose AUC responses and the first day of free-living cumulative glucose AUC. Because we will have repeated measures (4 days) of cumulative glucose AUC values in the field, mixed models will be used to assess the effects of in-lab glucose AUC on glucose responses to SB interruptions over 4 time points (day 1, 2, 3, and 4).

CONTACTS AND LOCATIONS:
Overall Officials: Britni R Belcher, PhD, MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California Keck School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to share IPD with other researchers outside of our study.